CLINICAL TRIAL: NCT02184312
Title: An Open-label, Non-randomised, Single-dose, Parallel-group Study of Pharmacokinetic Properties of 200 mg (2 x 100 mg Tablets Once Daily) and 300 mg (3 x 100 mg Tablets Once Daily) Nevirapine Extended Release Formulations Compared to 200 mg VIRAMUNE® Tablet as Well as to 400 mg Nevirapine Extended Release Tablet Following Oral Administration in Healthy Male Volunteers
Brief Title: Pharmacokinetic Properties of Two Dosages Nevirapine Extended Release (XR) Formulations Compared to VIRAMUNE® Tablet as Well as to Nevirapine XR Tablet in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1100.1517
Record Dates: First submitted 2014-07-08; First posted 2014-07-09 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
MeSH Terms: interventions — Nevirapine

ARMS (4):
- Nevirapine XR low dose (Experimental)
  Interventions: Drug: Nevirapine XR low dose
- Nevirapine XR medium dose (Experimental)
  Interventions: Drug: Nevirapine XR medium dose
- Nevirapine XR high dose (Active Comparator)
  Interventions: Drug: Nevirapine XR high dose
- Nevirapine (VIRAMUNE®) (Active Comparator): commercial product
  Interventions: Drug: Nevirapine (VIRAMUNE®)

INTERVENTIONS:
Drug: Nevirapine XR low dose
  Arms: Nevirapine XR low dose
Drug: Nevirapine XR medium dose
  Arms: Nevirapine XR medium dose
Drug: Nevirapine XR high dose
  Arms: Nevirapine XR high dose
Drug: Nevirapine (VIRAMUNE®)
  Arms: Nevirapine (VIRAMUNE®)

SUMMARY:
Study to determine the pharmacokinetic properties of 200 mg (2 x 100 mg tablets once daily) and 300 mg (3 x 100 mg tablets once daily) Nevirapine extended release formulations and to estimate relative bioavailability of these formulations as compared to 200 mg VIRAMUNE® tablet as well as to 400 mg Nevirapine extended release tablet

ELIGIBILITY:
Inclusion Criteria:

Healthy males according to the following criteria:

* Based upon a complete medical history, including the physical examination, vital signs (BP, PR), 12-lead ECG, clinical laboratory; values within normal ranges or deviating from normal without clinical relevance as considered by the investigator
* Values of Liver Function Test (LFT) have to be within normal ranges
* Age ≥18 and Age ≤60 years
* Body Mass Index (BMI) ≥18.5 and BMI ≤29.9 kg/m2
* Subjects must agree to minimize the risk of female partners becoming pregnant from the first dosing day until 3 months after the completion of the post study medical examination. Acceptable methods of contraception comprises barrier contraception and a medically accepted contraceptive method for the female partner (intra-uterine device with spermicide, hormonal contraceptive since at least two month)
* Signed and dated written informed consent prior to admission to the study in accordance with Good clinical practice (GCP) and the local legislation

Exclusion Criteria:

* Any finding of the medical examination (including BP, PR and ECG) deviating from normal and of clinical relevance
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders of clinical relevance
* Surgery of the gastrointestinal tract (except appendectomy and herniotomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
* Intake of drugs with a long half-life (>24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
* Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
* Participation in another trial with an investigational drug within two months prior to administration or during the trial
* Participation to trial BI 1100.1485 or any other intake of Nevirapine
* Smoker (>10 cigarettes or >3 cigars or >3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (more than 60 g/day)
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
* Excessive physical activities (within one week prior to administration or during the trial)
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 ms)
* A history of additional risk factors for Torsades des Pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)
* History of disease which affects the present situation
* Inability to understand the protocol requirements, instructions and study-related restrictions, the nature, scope, and possible consequences of the study
* Unlikely to comply with the protocol requirements, instructions and study-related restrictions; e.g., uncooperative attitude, inability to return for follow-up visits, and improbability of completing the study
* Subject is the investigator or any sub-investigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the study
* Vulnerable subjects (e.g. persons kept in detention)

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2008-04; Primary Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 144 hours after drug administration
Cmax (maximum measured concentration of the analyte in plasma) | up to 144 hours after drug administration

SECONDARY OUTCOMES:
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point) | up to 144 hours after drug administration
tmax (time from dosing to the maximum concentration of the analyte in plasma) | up to 144 hours after drug administration
λz (terminal rate constant in plasma) | up to 144 hours after drug administration
t1/2 (terminal half-life of the analyte in plasma) | up to 144 hours after drug administration
MRTpo (mean residence time of the analyte in the body after po administration) | up to 144 hours after drug administration
CL/F (apparent clearance of the analyte in the plasma after extravascular administration) | up to 144 hours after drug administration
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular dose) | up to 144 hours after drug administration
ka (absorption rate constant) | up to 144 hours after drug administration
Number of patients with adverse events | up to 36 days
Number of patients with abnormal changes in laboratory parameters | Screening, Day 1, 2, 3, 4, 5, 7, 15
Number of patients with clinically significant changes in vital signs (blood pressure (BP), pulse rate (PR)) | Screening, Day 1, 2, 15
Number of patients with clinically significant changes in 12-lead electrocardiogram (ECG) | Screening, Day 1, 15
Assessment of tolerability by investigator on a 4-point scale | up to 15 days after drug administration